CLINICAL TRIAL: NCT03313024
Title: Characterization of Immune Cell-trophoblast-interaction in Pregnancy Disorders
Brief Title: Berlin-Brandenburg Pregnancy Cohort
Acronym: BBPC
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Florian Herse, PhD, Charite University, Berlin, Germany
Other Study IDs: BBPC
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Preeclampsia; Pregnancy Complications; Diabetes Mellitus in Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the interplay of different immune cells and placental cells as well as their potential for the development of pregnancy complications. In particular, the translation of the uteroplacental syndrome into a maternal syndrome, considered in the multifactorial pregnancy disorder preeclampsia, will be investigated. Immune cell subtypes are causally involved in the formation and translation of preeclampsia by inducing an endothelial dysfunction which leads to cardiovascular damage.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women after giving informed consent
* pregnant with diagnosis of preeclampsia, gestational hypertension or gestational diabetes

Exclusion Criteria:

* infections
* alcohol and drug abuse
* manifest and chronic diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between 18 and 45 years of age without infections, severe or chronic diseases
Sampling Method: Probability Sample
Enrollment: 1580 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
T cell population content at the time of preeclampsia diagnosis compared to controls and verified by flow cytometry | at the time of preeclampsia diagnosis compared to controls at the same time point in pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Experimental and Clinical Research Center (ECRC), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided